CLINICAL TRIAL: NCT00992368
Title: Cost-effectiveness of Reduction Mammaplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, CARLOS DELANO MUNDIM ARAUJO, MD, PhD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1788.08
Record Dates: First submitted 2009-10-07; First posted 2009-10-09 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Breast,Hypertrophy; Cost-effectiveness
Keywords: Quality-Adjusted Life Years:A measurement index; Cost-Benefit Analysis:A method of comparing costs; Mammaplasty; QALY; Health-related quality of life; Cost-effectiveness; Breast
MeSH Terms: conditions — Gigantomastia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- reduction mammaplasty (Active Comparator): submitted to surgery
  Interventions: Procedure: reduction mammaplasty
- not reduction mammaplasty (No Intervention): not submitted to surgery

INTERVENTIONS:
Procedure: reduction mammaplasty — patients submitted to reduction mammaplasty
  Arms: reduction mammaplasty

SUMMARY:
Several works show breast hypertrophy as pain cause, postural alterations, dermatitis and decrease of the functional capacity and of the self-esteem. The economical evaluations are destined to esteem the costs in alternative ways of attendance to the health, comparing, for instance, clinical strategies with surgical strategies.

OBJECTIVE: To analyze cost-effectiveness in reduction mammaplasty.

DETAILED DESCRIPTION:
1. Design: This is a primary, prospective, analytical, controlled study in humans.
2. Settings: Data will be collected at the Plastic Surgery and Orthopedic and Traumatology Outpatient Clinics of the Samuel Libânio General Hospital (Hospital das Clínicas Samuel Libânio, HCSL), Pouso Alegre, MG, Brazil, in july/2008-december 2009.
3. Participants: Fifty women with breast hypertrophy (25 study group and 25 control group) according to the Sacchini index,12 aged 18 to 59 years, were consecutively selected to participate in this study.

   Pregnant women, and patients who gave birth or were breastfeeding less than one year before the beginning of the study, as well as patients with uncontrolled systemic diseases, acute diseases, breast asymmetry, who had undergone breast or spine surgery, and who had body-mass index (BMI) lower than 18.5 kg/m2 (low body weight) or greater than 30 kg/m2 (obese women) were excluded from the study.
4. Instruments: Pain intensity in the cervical, dorsal and lumbar regions of the back has been assessed using a visual analogue scale (VAS). also will be used SF36, HAQ 20 and SF-6D.

ELIGIBILITY:
Inclusion Criteria:

* Women with breast hypertrophy according to the Sacchini index

Exclusion Criteria:

* Pregnant women
* Patients who gave birth or were breastfeeding less than one year before the beginning of the study
* Patients with uncontrolled systemic diseases, acute diseases, or breast asymmetry
* Patients who had undergone breast or spine surgery
* Patients who had body-mass index (BMI) lower than 18.5 kg/m2 (low body weight) or greater than 30 kg/m2 (obese women)

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The total cost for procedure will be calculated with accuracy through the Brazilian software "TASY". To evaluate the effectiveness will be used the SHORT FORM 36, Visual Analogue Scale, Stanford Health Assessment Questionnaire 20 and SHORT FORM-6D | before the surgery (baseline)
The total cost for procedure will be calculated with accuracy through the Brazilian software "TASY". To evaluate the effectiveness will be used the SHORT FORM 36, Visual Analogue Scale, Stanford Health Assessment Questionnaire 20 and SHORT FORM-6D | 3 months after surgery
The total cost for procedure will be calculated with accuracy through the Brazilian software "TASY". To evaluate the effectiveness will be used the SHORT FORM 36, Visual Analogue Scale, Stanford Health Assessment Questionnaire 20 and SHORT FORM-6D | 6 months after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: CARLOS DM ARAUJO, MD, PhD, Principal Investigator — Federal University of São Paulo; DANIELA F VEIGA, MD, PhD, Study Director — Federal University of São Paulo; BERNARDO S HOCHMAN, MD, PhD, Study Director — Federal University of São Paulo; LUIZ EF ABLA, MD, PhD, Study Director — Federal University of São Paulo; LYDIA M FERREIRA, MD, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Carlos Dm Araujo, Pouso Alegre, Minas Gerais, Brazil

REFERENCES:
- [Result] Taylor AJ, Tate D, Brandberg Y, Blomqvist L. Cost-effectiveness of reduction mammaplasty. Int J Technol Assess Health Care. 2004 Summer;20(3):269-73. doi: 10.1017/s0266462304001072. PMID 15446755
- [Derived] Araujo CD, Veiga DF, Hochman BS, Abla LE, Oliveira AC, Novo NF, Veiga-Filho J, Ferreira LM. Cost-utility of reduction mammaplasty assessed for the Brazilian public health system. Aesthet Surg J. 2014 Nov;34(8):1198-204. doi: 10.1177/1090820X14539972. Epub 2014 Jun 27. PMID 24973340